CLINICAL TRIAL: NCT01925547
Title: Effect of Micellar Curcumin on Inflammation and Lipid Metabolism Markers
Brief Title: Micellar Curcumin and Metabolic Syndrome Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Jan Frank, Professor, Ph.D., University of Hohenheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0315679-HS3
Record Dates: First submitted 2013-07-23; First posted 2013-08-19 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Syndrome, Protection Against
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micellar curcumin (Experimental): Subjects receive three times per day four capsules of curcumin micelles. One capsule contains 20 mg of curcumin. At the beginning, after three and six weeks of intake, blood samples are collected.
  Interventions: Dietary Supplement: Micellar curcumin
- Placebo (Placebo Comparator): Subjects receive three times per day four capsules of placebo preparation. At the beginning, after three and six weeks of intake, blood samples are collected.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Micellar curcumin — 80 mg micellar curcumin (oral) three times a day for six weeks
  Arms: Micellar curcumin
Dietary Supplement: Placebo — Only the excipients (without curcumin) used to prepare the curcumin micelles are given as placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of micellar curcumin on inflammation and lipid metabolism markers in subjects at risk for the metabolic syndrome.

ELIGIBILITY:
Inclusion criteria:

* Total cholesterol > 5.2 mmol/L
* LDL cholesterol > 3.4 mmol/L
* Triglyceride > 2.26 mmol/L
* CRP > 2 mg/L

Exclusion criteria:

* Intake of drugs or dietary supplements
* Pregnant women and breastfeeding mothers
* Smokers
* Previous illnesses such as heart attack, cancer or dementia
* Addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) | At baseline and 6 weeks
  Serum CRP in mg/L

SECONDARY OUTCOMES:
Plasma curcumin concentrations | At baseline and 6 weeks
  Concentrations (in nmol/L) of curcumin and curcumin conjugates in plasma
Serum alanine transaminase activity | At baseline and 6 weeks
  Serum activity of ALT in U/L
Fasting blood glucose | At baseline and 6 weeks
  Fasting blood glucose in mmol/L
Plasma tumor necrosis factor alpha | At baseline and 6 weeks
  Plasma concentrations of TNFα in pg/mL
Serum uric acid | At baseline and 6 weeks
  Serum concentrations of uric acid in g/L
Plasma albumin | At baseline and 6 weeks
  Plasma concentrations of albumin in g/L
Serum total cholesterol | At baseline and 6 weeks
  Serum total cholesterol in mmol/L
Serum triacylglycerols | At baseline and 6 weeks
  Serum triacylglycerols in mmol/L
Serum HDL cholesterol | At baseline and 6 weeks
  Serum HDL cholesterol in mmol/L
Serum LDL cholesterol | At baseline and 6 weeks
  Serum LDL cholesterol in mmol/L
Serum aspartate transaminase activity | At baseline and 6 weeks
  Serum activity of AST in U/L
Serum gamma glutamyl transferase activity | At baseline and 6 weeks
  Serum activity of gamma-GT in U/L
Serum alkaline phosphatase activity | At baseline and 6 weeks
  Serum activity of ALP in U/L
Serum bilirubin | At baseline and 6 weeks
  Serum concentrations of bilirubin in g/L
Plasma interleukine 6 | At baseline and 6 weeks
  Plasma concentrations of IL-6 in pg/mL
Serum insulin | At baseline and 6 weeks
  Serum concentrations of insulin in pg/mL
Body weight | At baseline and 6 weeks
  Body weight in kg
Diastolic blood pressure | At baseline and 6 weeks
  Diastolic blood pressure in mmHg
Serum creatinine | At baseline and 6 weeks
  Serum concentrations of creatinine in g/L
Systolic blood pressure | At baseline and 6 weeks
  Systolic blood pressure in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Ph.D., Principal Investigator — University of Hohenheim
Locations (1):
- Institute of Biological Chemistry and Nutrition, University of Hohenheim, Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Kocher A, Bohnert L, Schiborr C, Frank J. Highly bioavailable micellar curcuminoids accumulate in blood, are safe and do not reduce blood lipids and inflammation markers in moderately hyperlipidemic individuals. Mol Nutr Food Res. 2016 Jul;60(7):1555-63. doi: 10.1002/mnfr.201501034. Epub 2016 May 23. PMID 26909743